CLINICAL TRIAL: NCT03080519
Title: A Multicenter Registry of Endovascular Therapy for Renal Artery Stenosis in China
Brief Title: Endovascular Therapy for Renal Artery Stenosis in China
Acronym: ETRAS-China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Xiongjing Jiang, Professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-ZX-0214
Record Dates: First submitted 2017-03-02; First posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Renal Artery Obstruction; Hypertension, Renovascular
Keywords: renal artery stenosis; balloon angioplasty; stents
MeSH Terms: conditions — Renal Artery Obstruction; Hypertension, Renovascular

STUDY DESIGN:
Intervention Model Description: Intervational Therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endovascular Therapy (Experimental): Renal artery revascularization
  Interventions: Procedure: Endovascular Therapy

INTERVENTIONS:
Procedure: Endovascular Therapy — Balloon angioplasty and stenting for renal artery stenosis

SUMMARY:
A multicenter prospective registry planned to recruit more than 5 000 patients with renal artery stenosis was carried out in China. This primary purpose of this study was to evaluate the safety and efficacy of renal artery revascularization in the real world. The secondary purpose was to investigate the etiologic distribution of renal artery stenosis and optimize the indications for renal artery revascularization.

DETAILED DESCRIPTION:
Currently,the endovascular therapy of renal artery stenosis (especially atherosclerotic) remains in dispute. Some randomized control trials published in recent years (including ASTRAL and CORAL trials) showed the lack of additional benefit for renal artery revascularization compared with sole medical therapy. However,these randomized control trials presented a number of limitations including low numbers of patients and non-stringent inclusion criteria. Given clinical medical practice entering the era of big data, the large-sample real-word studies would be more objective to answer some pending issues of randomized controlled trial.Therefore,a multicenter prospective registry planned to recruit more than 5 000 patients with renal artery stenosis was carried out. This primary purpose of this study was to evaluate the safety and efficacy of renal artery revascularization in the real world. The secondary purpose was to investigate the etiologic distribution of renal artery stenosis and optimize the indications for renal artery revascularization.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 14 at the time of informed consent
2. Diameter reduction of renal artery or main branch of renal artery≥ 60%,and ≥2 of four following conditions met:1)systolic hyperemic pressure gradient >20 mm Hg,2)captopril renoscitigraphy positive in the lesion side

   ,3)renin-angiotensin-aldosterone system significantly activated and 4)severe reduction (>25%) of glomendar filtration rate in the lesion side
3. office systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg while receiving 3 antihypertensive drugs,or office systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg without antihypertensive drugs
4. Serum creatinine level<264umol/L
5. Length of ipsilateral kidney ≥7.0 cm and glomendar filtration rate ≥10 ml／min
6. Urine protein <2+

Exclusion Criteria:

1. Unable to provide informed consent
2. Unstable condition and unable to tolerate interventional therapy
3. intolerance to antiplatelet drugs or contrast medium
4. vascular anatomy not suitable for endovascular therapy
5. Pregnant, nursing, or planning to be pregnant

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Efficacy：Change in blood pressure compared to baseline | Measured at 1 month and every 6 months thereafter from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
Safety: Change in estimated glomerular filtration rate compared to baseline | Measured at 1 month and every 6 months thereafter from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months

SECONDARY OUTCOMES:
Device or procedure related acute adverse events (renal artery dissection,renal artery perforation,bleeding,and etc.) | Perioperative period
The incidence of major adverse event (cardiovascular or renal death,myocardial infarction,hospitalization for congestive heart failure, stroke, and renal failure) | Measured at 1 month and every 6 months thereafter from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
The incidence of renal artery restenosis(>50%) | Measured every 6 months from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiongjing Jiang, Dr., Principal Investigator — Fuwai Hospital, National Center for Cardiovascular Disease, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (16):
- China (16):
  - Beijing Renhe Hospital, Beijing, Beijing Municipality
  - Fuwai Hospital, National Center for Cardiovascular Disease, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - Daping Hospital, Chongqing, Chongqing Municipality
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Guangdong General Hospital, Guangzhou, Guangdong
  - The Eighth Affiliated Hospital of Sun Yat-sen University, Shenzhen, Guangdong
  - Hongqi Hospital, Mudanjiang, Heilongjiang
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The General Hospital of Shenyang Military, Shenyang, Liaoning
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Xi'an NO.3 Hospital, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Zhejiang Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No